CLINICAL TRIAL: NCT01458483
Title: Acute Carotid Sinus Endovascular Stimulation II Study
Acronym: ACES II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACES II
Record Dates: First submitted 2011-08-25; First posted 2011-10-24 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baroreceptor Stimulation (Experimental)
  Interventions: Device: Baroreceptor Stimulation

INTERVENTIONS:
Device: Baroreceptor Stimulation — The stimulation catheter may be placed in different locations within the IJV at the level of the cervical spine vertebrae. Stimulation amplitudes will be varied from 0.1 mA to 20 mA.

SUMMARY:
The Acute Carotid Sinus Endovascular Stimulation II (ACES II) Study is a multicenter, prospective, non-randomized study that is being conducted to evaluate the feasibility of endovascular stimulation of carotid sinus nerves via an electrophysiology (EP) catheter advanced into the internal jugular vein (IJV). The current study investigates the hypothesis that intraoperative electrical stimulation of the carotid sinus from the IJV will result in an acute and dose-dependent reduction in blood pressure and heart rate.

DETAILED DESCRIPTION:
All study objectives are being assessed during the intraoperative baroreceptor stimulation. No subsequent testing will be performed. The follow-up visit is only intended to assess for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old
* Subject is hypertensive (defined as at least one in-office Systolic BP measurement ≥140 mm Hg or Diastolic BP ≥90 mm Hg within three months prior to enrollment
* Subject is undergoing a cardiac catheterization involving right heart catheterization and/or EP procedures.
* Subject (or subject's legally authorized representative) is able and wiling to give informed consent

Exclusion Criteria:

* Subject has an ejection fraction (EF) less than 35% (by most recent echocardiography in the past 6 months) and there has been no change in clinical status relative to EF
* Subject is a woman who is pregnant, nursing, or of child bearing potential and is not on a reliable form of birth control
* Subject is enrolled or is planning to participate in a concurrent drug and/or device study during the course of this clinical trial. Co-enrollment in concurrent trials is only allowed with documented pre-approval from the Medtronic study manager, documenting that there is not a concern that co-enrollment could confound the results of this trial.
* Subject is unable or unwilling to participate with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure during electrical stimulation | Intraoperative testing only
Change in diastolic blood pressure during electrical stimulation | Intraoperative testing only

SECONDARY OUTCOMES:
Characterize number and type of side effects seen during stimulation | Intraoperative testing only

CONTACTS AND LOCATIONS:
Overall Officials: Randy Lieberman, M.D., Principal Investigator — Harper Hospital
Locations (1):
- Detroit, Michigan, United States

REFERENCES:
- See also: Related Info — http://www.nlm.nih.gov/medlineplus/highbloodpressure.html